CLINICAL TRIAL: NCT02848729
Title: A Randomized, 2-Way, Parallel, Single-Blind Pharmacokinetic Study to Evaluate the Interaction Between Intravenous Morphine and Orally or Intravenously Administered Acetaminophen in Healthy Subjects
Brief Title: Drug Interactions Between Morphine and Orally or IV Administered Acetaminophen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MNK14564059
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: Post-surgical pain; Pharmacokinetics
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Acetaminophen; Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: Oral Acetaminophen (Experimental): Treatment A = 4 repeat doses of 1,000 mg oral acetaminophen (2 x 500 mg tablets) and an IV infusion of saline every 6 hours (Hours -6, 0, 6, and 12), and 2 infusions of intravenous (IV) morphine (0.125 mg/kg) at Hours 0 and 6
  Interventions: Drug: Oral Acetaminophen; Drug: IV Morphine; Drug: Saline
- Treatment B: IV Acetaminophen (Experimental): Treatment B = 4 repeat doses of IV acetaminophen (1,000 mg/100 mL) and 2 placebo tablets every 6 hours (Hours -6, 0, 6, and 12), and 2 infusions of IV morphine (0.125 mg/kg) at Hours 0 and 6.
  Interventions: Drug: IV Acetaminophen; Drug: IV Morphine; Drug: Placebo Tablets

INTERVENTIONS:
Drug: Oral Acetaminophen — Acetaminophen for oral administration (2 tablets, 500 mg/tablet)
  Other Names: APAP Oral
  Arms: Treatment A: Oral Acetaminophen
Drug: IV Acetaminophen — Acetaminophen for intravenous (IV) administration (1,000 mg/100 mL)
  Other Names: APAP IV
  Arms: Treatment B: IV Acetaminophen
Drug: IV Morphine — Morphine for IV administration (0.125 mg/kg)
Drug: Placebo Tablets — Placebo tablets matching oral acetaminophen
  Arms: Treatment B: IV Acetaminophen
Drug: Saline — Saline placebo matching IV acetaminophen
  Arms: Treatment A: Oral Acetaminophen

SUMMARY:
Morphine is the opioid used to treat pain after surgery. Acetaminophen (called APAP) can reduce the amount of opioids needed for this.

The problem is that morphine slows down digestion. That can delay pain relief from APAP pills. It can even change what the body does to the drug [pharmacokinetics (PK)].

Some doctors have started using intravenous (IV) APAP with morphine, instead of the pills.

This study will measure the PK of APAP pills and IV when used with morphine in healthy volunteers.

IV APAP will likely be more effective and cause fewer side effects when used with morphine to treat pain after surgery.

DETAILED DESCRIPTION:
Acetaminophen can significantly reduce the use of opioid analgesics when both are used concomitantly for treating moderate to severe pain. The use of IV acetaminophen used concomitantly with opioids has increased in practice for postsurgical pain relief over orally administered acetaminophen because it provides an immediate peak plasma concentration and is believed to provide a faster analgesic effect. Opioids used to treat pain inhibit gastrointestinal motility, including delaying gastric emptying. In patients receiving opioids the absorption of orally administered acetaminophen may be delayed and could result in gastric accumulation of acetaminophen thereby markedly changing the pharmacokinetic profile. The opioid-induced inhibition of gastrointestinal motility would not be expected to affect IV acetaminophen pharmacokinetics. Thus coadministered IV acetaminophen with opioid would yield better outcome in efficacy and reduced risk of side effects comparing with coadministration of oral acetaminophen and opioids.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a health status of "healthy" assessed by the investigator and defined as no clinically significant deviation from normal medical history, physical examination, vital signs, and clinical laboratory determinations.
2. Subject must have a body mass index ≥ 19.0 and ≤ 32.0 kg/m² with a minimum weight of 110 pounds (50 kg) at Screening.

Exclusion Criteria:

1. Subject has a positive test result for human immunodeficiency virus (HIV), hepatitis B (surface antigen), or hepatitis C virus antibody at screening.
2. Subject has a history of any drug allergy, hypersensitivity, or intolerance to acetaminophen or morphine/opioids or to any of the excipients in the IV or oral formulations used.
3. Subject has an oxygen saturation of less than 95% while awake at screening and check-in.
4. Subject has a positive test result for drugs of abuse (minimum: opioids, barbiturates, cannabinoids, benzodiazepines, cocaine, amphetamine) or alcohol at the screening and check-in.
5. Subject has donated or had significant loss of whole blood (480 mL or more) within 30 days, or plasma within 14 days prior to dosing.
6. Subject has any other medical, psychiatric and/or social reason for exclusion as determined by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (3):
- United States (3):
  - University of Arizona College of Pharmacy, Tucson, Arizona
  - NEMA Research, Inc., Naples, Florida
  - The University of Rhode Island College of Pharmacy, Kingston, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raffa RB, Pawasauskas J, Pergolizzi JV Jr, Lu L, Chen Y, Wu S, Jarrett B, Fain R, Hill L, Devarakonda K. Pharmacokinetics of Oral and Intravenous Paracetamol (Acetaminophen) When Co-Administered with Intravenous Morphine in Healthy Adult Subjects. Clin Drug Investig. 2018 Mar;38(3):259-268. doi: 10.1007/s40261-017-0610-4. PMID 29214506

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Acetaminophen: Treatment A = 4 repeat doses of 1,000 mg oral acetaminophen (2 x 500 mg tablets) and an intravenous (IV) infusion of saline every 6 hours (Hours -6, 0, 6, and 12), and 2 infusions of IV morphine (0.125 mg/kg) at Hours 0 and 6.
- IV Acetaminophen: Treatment B = 4 repeat doses of IV acetaminophen (1,000 mg/100 mL) and 2 placebo tablets every 6 hours (Hours -6, 0, 6, and 12), and 2 infusions of IV morphine (0.125 mg/kg) at Hours 0 and 6.
Period: Overall Study
Arm/Group | Oral Acetaminophen | IV Acetaminophen
Started | 27 | 23
Per Protocol Population | 11 | 11
Safety Population | 27 | 23
Completed | 11 | 12
Not Completed | 16 | 11
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Emesis | 15 | 11

BASELINE CHARACTERISTICS:
Population: All participants with emesis were removed from the study, with no replacement. Because 7 of 9 females had emesis at the first dose, an amendment was written to exclude females. Therefore, demographics are provided for the per protocol population.
Groups:
- Oral Acetaminophen: Treatment A = 4 repeat doses of 1,000 mg oral acetaminophen (2 x 500 mg tablets) and an IV infusion of saline every 6 hours (Hours -6, 0, 6, and 12), and 2 infusions of IV morphine (0.125 mg/kg) at Hours 0 and 6.
- Total: Total of all reporting groups
Arm/Group | Oral Acetaminophen | IV Acetaminophen | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (9.82) | 32.5 (11.25) | 32.8 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 9 | 16
  Black or African American | 2 | 2 | 4
  Hispanic or Latino Ethnicity | 4 | 6 | 10
  Not Hispanic or Latino | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve Over 6 Hours (AUC6) for Acetaminophen
Description: The area under the plasma drug concentration-time curve (AUC) is an estimate of how much drug remains available for the body to use, within a certain amount of time after the drug is administered. AUC6 is reported for each of the 6-hour dosing periods of acetaminophen before (hours -6 to 0), during (hours 0-6 and 6-12) and after (hours 12-18) morphine co-administration for each route of acetaminophen administration
Time Frame: hours -6 to 0, 0-6, 6-12, and 12-18 during treatment with each mode of acetaminophen administration
Population: Per-protocol population, which is defined as the participants who received all study medication, provided all 33 blood samples within required time points and completed the study with no major protocol deviations.
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter (h*mcg/mL)
Groups:
- First Dose - Before Morphine Co-administration: AUC6 for acetaminophen before morphine co-administration (hours -6 to -1)
- Second Dose - During Morphine Co-administration: AUC6 for acetaminophen during morphine co-administration (hours 0 to 6)
- Third Dose - During Morphine Co-administration: AUC6 for acetaminophen during morphine co-administration (hours 6 to 12)
- Fourth Dose - After Morphine Co-administration: AUC6 for acetaminophen after morphine co-administration (hours 12 to 18)
Arm/Group | First Dose - Before Morphine Co-administration | Second Dose - During Morphine Co-administration | Third Dose - During Morphine Co-administration | Fourth Dose - After Morphine Co-administration
Number analyzed (Participants) | 11 | 11 | 11 | 11
hour*microgram per milliliter (h*mcg/mL)
  Treatment A: Oral Acetaminophen | 31.00 (5.11) | 28.51 (5.96) | 25.31 (11.59) | 52.38 (13.48)
  Treatment B: IV Acetaminophen | 42.56 (3.94) | 44.37 (4.46) | 43.59 (4.21) | 49.05 (3.95)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve Over 18 Hours (AUC18) for Acetaminophen After First Morphine Co-administration
Description: AUC18 is reported for the 18-hour treatment period after first morphine co-administration, for each route of acetaminophen administration
Time Frame: hours 0-18 during treatment with each mode of acetaminophen administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter (h*mcg/mL)
Groups:
- After First Dose of Morphine Co-administration: AUC18 after first dose of morphine co-administration (hours 0-18)
Arm/Group | After First Dose of Morphine Co-administration
Number analyzed (Participants) | 11
hour*microgram per milliliter (h*mcg/mL)
  Treatment A: Oral Acetaminophen | 82.50 (23.28)
  Treatment B: IV Acetaminophen | 63.58 (6.74)

3. Primary Outcome: Maximum Concentration (Cmax) of Acetaminophen
Description: Following the administration of drugs, the plasma concentration generally reaches a single, well-defined peak which is the most drug that is available for the body to use (Cmax). Cmax is reported for the 6-hour dosing periods before (hours -6 to 0), during (hours 0-6 and 6-12), and after (hours 12-18) morphine co-administration for each route of acetaminophen administration.
Time Frame: hours -6 to 0, 0-6, 6-12, and 12-18 during treatment with each mode of acetaminophen administration
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- First Dose - Before Morphine Co-administration: Pharmacokinetics of oral acetaminophen before morphine co-administration (hours -6 to -1)
- Second Dose - During Morphine Co-administration: Pharmacokinetics of oral acetaminophen during morphine co-administration (hours 0 to 6)
- Third Dose - During Morphine Co-administration: Pharmacokinetics of oral acetaminophen during morphine co-administration (hours 6 to 12)
- Fourth Dose - After Morphine Co-administration: Pharmacokinetics of oral acetaminophen during morphine co-administration (hours 12 to 18)
Arm/Group | First Dose - Before Morphine Co-administration | Second Dose - During Morphine Co-administration | Third Dose - During Morphine Co-administration | Fourth Dose - After Morphine Co-administration
Number analyzed (Participants) | 11 | 11 | 11 | 11
mcg/mL
  Treatment A: Oral Acetaminophen | 11.6 (4.11) | 7.29 (1.82) | 7.25 (3.95) | 13.5 (3.31)
  Treatment B: IV Acetaminophen | 22.6 (3.83) | 17.0 (1.48) | 17.5 (1.93) | 28.5 (4.31)

4. Primary Outcome: Time to Maximum Concentration (Tmax) of Acetaminophen
Description: Following the administration of drugs, the time at which the plasma concentration reaches Cmax is called Tmax. Tmax is reported for the 6-hour dosing periods before (hours -6 to 0), during (hours 0-6 and 6-12) and after (hours 12-18) morphine co-administration for each route of acetaminophen administration.
Time Frame: hours -6 to 0, 0-6, 6-12 and 12-18 during treatment with each mode of acetaminophen administration
Population: Per-protocol population
Measure: Mean (Full Range); unit: hours
Arm/Group | First Dose - Before Morphine Co-administration | Second Dose - During Morphine Co-administration | Third Dose - During Morphine Co-administration | Fourth Dose - After Morphine Co-administration
Number analyzed (Participants) | 11 | 11 | 11 | 11
hours
  Oral Acetaminophen | 1.48 [0.75 to 2.02] | 1.64 [0.50 to 3.00] | 3.26 [0.50 to 5.85] | 2.84 [1.17 to 4.02]
  IV Acetaminophen | 0.25 [0.25 to 0.27] | 0.50 [0.50 to 0.50] | 0.51 [0.50 to 0.57] | 0.25 [0.25 to 0.28]

ADVERSE EVENTS:
Time Frame: From start of the study to the end of study (approximately 2 weeks, including wash-out period)
Description: The safety analysis set, defined as all participants who received study drug, was used for the adverse events module.
Arm/Group | Oral Acetaminophen | IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 22/27 | 17/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Acetaminophen (N=27) | IV Acetaminophen (N=23)
Vomiting (Gastrointestinal disorders) | 15 | 11
Nausea (Gastrointestinal disorders) | 12 | 10
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 4
Somnolence (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 2
Asthenia (General disorders) | 2 | 0
Catheter site pain (General disorders) | 2 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Feeling of relaxation (General disorders) | 1 | 0
Infusion site pruritus (General disorders) | 0 | 1
Euphoric mood (Psychiatric disorders) | 1 | 3
Irritability (Psychiatric disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Micturition disorder (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No